CLINICAL TRIAL: NCT02067546
Title: Innovative Toilet Seat Test for Patients With Symptoms of Constipation and/or Emptying Disorders
Acronym: constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-13-RY-244-CTIL
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Constipation
Keywords: constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental toilet seat (Experimental): Experimental toilet seat for 1 month
  Interventions: Device: Experimental toilet seat
- Standard toilet seat (Sham Comparator): Standard toilet seat for 1 month
  Interventions: Device: Standard toilet seat

INTERVENTIONS:
Device: Experimental toilet seat
  Arms: Experimental toilet seat
Device: Standard toilet seat
  Arms: Standard toilet seat

SUMMARY:
Emptying disorders are of the most common causes of constipation. An adjustable toilet seat was designed by " Shva-Nach" Ltd company, and is designed to facilitate the angle sitting position.

Its efficacy will be evaluated in the current study, on 50 volunteers who suffer from constipation and meet the Rome 3 criteria for constipation.

DETAILED DESCRIPTION:
Emptying disorders are of the most common causes of constipation. Laxatives are usually unsuccessful. Behavioral therapy such as anorectal biofeedback , have a limited success in most hospitals in this country. Toilet seat that lifts the legs and brings us into a sitting position closer to squatting (which is the desired physiological position) can relieve these patients in the emptying process.

The Company " Shva-Nach" Ltd. and its design team designed a seat at an angle slightly elevated and a toilet stool customized to the personal anatomy of each subject.

The purpose of the study: evaluating efficacy elevated toilet seat with a support of a brackets stool making emptying easier in patients with constipation and difficulty in emptying.

Methods: An open, randomized, crossover study in use of a toilet seat and comparing it to a standard seat.

ELIGIBILITY:
Inclusion criteria:

1. Patients suffering from constipation and meet the criteria of Rome 3. No sub - distribution by emptying disorders or decreased stool frequency
2. Age group 18-80 years
3. Study population may include patients suffering from metabolic diseases such as diabetes mellitus, hypothyroidism and hypercalcemia.
4. Patients who understand the goals of the research and collaborate

Exclusion Criteria:

1. Patients who do not understand the goals of the research and / or unable to cooperate.
2. women with known pregnancy - second trimester and up
3. Patients with obesity - BMI> 35 and / or weight over 120 kg
4. Neurological diseases - dementia, Parkinson's disease, CVA, multiple sclerosis, muscular dystrophy, spinal cord injury
5. Disabled patients on wheelchairs.
6. Patients with active anal fissure / fistula, active inflammation of the colon, patients after resection of the colon.
7. Minors and no judgment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in bowel movement frequency | 2 months

SECONDARY OUTCOMES:
Improvement in quality of life | 2 months
  According to QOL questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel, Israel